CLINICAL TRIAL: NCT01773460
Title: A Multicenter Randomized, Double Blind, Placebo- Controlled, Phase II Study to Compare Endocrine Treatment Alone Versus Endocrine Treatment With Everolimus in Patients With HR+/HER2- Metastatic Breast Cancer and Progression After Previous Treatment With Exemestane and Everolimus
Brief Title: Everolimus Beyond Progress for Patients Who Had Progress Under Everolimus and Exemestane
Acronym: Evelyn
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was stopped terminated early due to low recruitment.
Sponsor: GBG Forschungs GmbH (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GBG 76
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Breast Cancer
Keywords: everolimus progress exemestane; treated with exemestane and everolimus; progress under this treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (Experimental): Everolimus is given beyond progress
  Interventions: Drug: Everolimus
- Everolimus-placebo (Placebo Comparator): Everolimus-placebo is given beyond progress
  Interventions: Drug: Everolimus-placebo

INTERVENTIONS:
Drug: Everolimus — Everolimus is given beyond progress (comparison with placebo)
  Other Names: Everolimus, Afinitor, RAD-001
  Arms: Everolimus
Drug: Everolimus-placebo — Everolimus-placebo
  Other Names: placebo
  Arms: Everolimus-placebo

SUMMARY:
Everolimus will be given to patients with metastatic breast cancer who already has a progress taking Everolimus but with a change in the endocrine treatment.

DETAILED DESCRIPTION:
With continuation of endocrine treatment of breast cancer an adaptive upregulation of different signaling cascades including the PI3K/akt/mTOR pathway results in cell growth stimulation and results in resistance to endocrine therapies. One way to restore endocrine sensitivity is the inhibition of the mTOR pathway in combination with endocrine therapy leading to an increase in PFS compared with endocrine therapy alone. Guidelines recommend the sequential treatment with different endocrine therapies. It therefore appears reasonable to explore if sensitivity can be restored by changing the subsequent endocrine combination partner of Everolimus in case of failure of a combined endocrine-everolimus therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements.

  2. Complete baseline documentation must be submitted via the web-based data collection system MedCODES® to the GBG Forschungs GmbH.

  3. Histological confirmed hormone receptor positive (HR+); HER2-negative carcinoma of the breast. Every effort should be made to make paraffin embedded tissue or slides from the original tumor and/or from metastatic tissue available for confirmation of diagnosis and additional translational research.

  4. Postmenopausal women 5. HER2-negative, hormone-receptor-positive, locally advanced or metastatic stage of disease not amenable to curative treatment by surgery or radiotherapy alone.

  6. No indication for chemotherapy 7. Patients must have either measurable or non-measurable target lesions according to RECIST criteria. Complete staging work-up within 4 weeks prior to registration including chest and abdominal CT scan or MRI (exceptionally chest X-ray and abdominal ultrasound), and bone scan. Further tests have to be performed according to RECIST or as clinically indicated.

  8. Disease progression during or after previous exemestane and everolimus treatment as follows (everolimus has to be given previously for at least 12 weeks, treatment-free interval of everolimus for a maximum of 6 weeks until randomization) 9. The following previous systemic treatments are eligible:
* Previous participation in other everolimus-containing trials, e.g. the GeparQuinto, BOLERO, 4EVER study is allowed.
* (Neo)Adjuvant and up to 1 chemotherapy regimen for metastatic breast cancer
* Maximum of two lines as palliative endocrine monotherapy
* Treatment with bisphosphonates and/or denosumab (adjuvant and/or palliative) 10. At least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation field or there must be pathologic proof of newly progressive disease.

  11. Age ≥ 18 years 12. ECOG performance status 0-2 13. Laboratory requirements:
  * Absolute neutrophil count at least 1500 cells/microliter,
  * hemoglobin ≥9.0 g/dL (hemoglobin <9.0 g/dL is acceptable if it is corrected by growth factor or transfusion)
  * platelet count at least 100,000 cells/microliter.
  * bilirubin at least 1.5x the upper limit of normal for the institution (ULN);
  * elevation of transaminases and alkaline phosphatase <3x ULN or <5x ULN for patients with liver metastases.
  * BUN (blood urea nitrogen) ≤ULN
  * Fasting plasma glucose (FPG) ≤160 mg/dL or ≤8.9 mmol/L
  * Fasting serum cholesterol ≤ 300mg/dl or 7.75mmol/L (LDL cholesterol <190mg/dl) and fasting triglyceride ≤2.5xULN (<300mg/dl). In case one or both of these thresholds are exceeded the patient can only be included after initiation of a statin therapy and when above mentioned values have been achieved.

INR ≤2.0 Creatinine not more than 2.0 x ULN or creatinine-clearance >40 ml/min (according to Cockcroft-Gault).

Urine dipstick for proteinuria <2+. Patients discovered to have ≥2+ proteinuria on dipstick urinalysis should undergo a 24 hour urine collection and must demonstrate ≤1 g of protein in 24 hours 14. Patients must be available and compliant for treatment and follow-up. Patients registered on this trial must be treated and followed up at the participating or a cooperating center.

Exclusion Criteria:

* 1. No documented progression on everolimus plus exemestane 2. Known hypersensitivity reaction to the compounds or incorporated substances 3. Treatment with medroxyprogesteronacetate, megestrolacetate, or high-dose estradiol within 12 weeks of study entry.

  4. Concurrent immunotherapy or hormonal therapy (contraceptive and/or replacement therapy). Bisphosphonates or denosumab may be continued 5. Life expectancy of less than 3 months. 6. Parenchymal brain metastases, unless adequately controlled by surgery and/or radiotherapy.

  7. Any ongoing toxicity from prior anti-cancer therapy that is grade 3-4 and/or that is progressing in severity, except alopecia or anemia controlled by growth factors.

  8. Any previous adverse event grade 3-4 or serious adverse event during treatment with exemestane and everolimus which led to treatment discontinuation 9. Known or suspected congestive heart failure (>NYHA I) and/or coronary heart disease, angina pectoris requiring anti-anginal medication, previous history of myocardial infarction ≤ 6months, evidence of transmural infarction on ECG, un- or poorly controlled arterial hypertension (i.e. BP >150/100 mmHg under treatment with two antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease 10. Currently active infection 11. History of other malignancies within the last 5 years which significantly affect the diagnosis, assessment or prognosis of metastatic breast cancer.

  12. Malabsorption syndrome or insufficient gastrointestinal function, preexisting diagnosis of ulcerative colitis 13. Concurrent treatment with other experimental drugs; participation in another clinical trial with any investigational not marketed drug within 30 days prior to study entry.

  14. Insufficiently controlled diabetes 15. known HIV infection or chronic hepatitis B or C 16. seriously impaired liver function (Child-Pugh, class C) 17. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures (including severe pulmonary conditions, AIDS and serious active infection and diabetes mellitus).

  18. Male patients 19. Known HIV infection or chronic or history of hepatitis B or C 20. Seriously impaired liver function (Child-Pugh, class C)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
progression free survival | 3 years
  comparison of progression free survival between the two arms: with Everolimus or with Everolimus-placebo

SECONDARY OUTCOMES:
overall survival | 3 years
  comparison of the overall survival between the 2 arms
clinical benefit Rate(CBR) | 3 years
  Clinical Benefit Rate (CBR) is defined as all patients with a complete, partial response and stable disease for at least 24 weeks
chemo-free interval | 3 years
  chemo-free interval is defined as time from last day of chemotherapy in the metastatic setting until first day of next chemotherapy or in patients who have not received chemotherapy in the metastatic setting: the first diagnosis of metastases until start of 1st-line chemotherapy in the metastatic setting.
safety by toxicity | 3 years
  Safety by toxicity grades is defined by the NCI-CTCAE version 4.03
compliance | 3 years
  Compliance will be assessed by the number and reasons of patients whose treatment had to be reduced, delayed or permanently stopped
biological marker | starting in 3 years, biomaterial will be stored, later research possible
  Bone marker estimation in blood and/or urine

OTHER OUTCOMES:
translational research: search for markers for prediction | starting in 3 years, biomaterial will be stored, later research possible
  PI3K/mTor and other related markers in tissue collected directly before study entry

CONTACTS AND LOCATIONS:
Overall Officials: Sibylle Loibl, Prof., Study Chair — Krankenhaus Offenbach
Locations (1):
- Klinikum Offenbach, Offenbach, Hesse, Germany